CLINICAL TRIAL: NCT01751646
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Effectiveness of Vitamin D3 50,000 IU Every 4 Weeks to Increase Bone Mineral Density and Decrease Tenofovir-Induced Hyperparathyroidism in Youth With HIV Infection Being Treated With Tenofovir-Containing Combination Antiretroviral Therapy (cART)
Brief Title: Vitamin D Absorption in HIV Infected Young Adults Being Treated With Tenofovir Containing cART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ATN 109 Version 2.0
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2018-11

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Vitamin D3 50,000 IU (Experimental): Subjects randomized to Group A will receive Vitamin D3 50,000 IU orally every four weeks by directly observed therapy (DOT). In addition all subjects receive a multivitamin (MVI) that contains ingredients not to exceed 600 IU of vitamin D3 and 200 mg of Calcium (Ca). Subjects will self-administer one MVI tablet orally once daily.
  Interventions: Dietary Supplement: Vitamin D3 50,000 IU
- Group B: Vitamin D3 placebo (Placebo Comparator): Subjects randomized to Group B will receive Vitamin D3 placebo orally every four weeks by DOT. In addition all subjects receive a MVI that contains ingredients not to exceed 600 IU of vitamin D3 and 200 mg of Ca. Subjects will self-administer one MVI tablet orally once daily.
  Interventions: Dietary Supplement: Vitamin D3 placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 50,000 IU — Group A: Vitamin D3 50,000 IU orally every four weeks by DOT
  Other Names: Vitamin D3
  Arms: Group A: Vitamin D3 50,000 IU
Dietary Supplement: Vitamin D3 placebo — Group B: Vitamin D3 placebo orally every four weeks by DOT
  Other Names: Placebo
  Arms: Group B: Vitamin D3 placebo

SUMMARY:
This is a 48 week randomized double-blind, placebo-controlled prospective cohort study of adolescents and young adults with HIV infection in the Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) who are currently being treated with cART that includes tenofovir disoproxil fumarate (TDF) as one component of the regimen that includes at least three Food and Drug Administration (FDA)-approved antiretroviral (ARV) drugs for at least 180 days.

DETAILED DESCRIPTION:
This is a 48 week randomized double-blind, placebo-controlled prospective cohort study of adolescents and young adults with HIV infection in the ATN who are currently being treated with cART that includes TDF as one component of the regimen that includes at least three Food and Drug Administration (FDA)-approved ARVs for at least 180 days. Subjects must have at least one documented viral load that is below 200 copies/mL that is collected following initiation of TDF containing cART and greater than 90 days prior to randomization; no viral load above 200 copies/mL if measured within the 90 days prior to randomization; and an HIV viral load obtained at screening that is below 200 copies/mL.

Treatment assignments will be balanced by subject sex at birth, age (<20 years vs. >=20 years), and race (African American vs. other). Enrolled subjects will be randomized to receive vitamin D3 50000 IU or matching placebo, given orally every four weeks by DOT. In addition to the randomized study agent, all subjects will receive a MVI to be taken orally once daily. This "standard" MVI will contain ingredients not to exceed 600 IU of vitamin D3 and 200 mg Ca.

Dual energy x-ray absorptiometry (DXA) measurement of bone mineral content (BMC)/bone mineral density (BMD) of whole body, spine, and hip, will be performed at baseline and study weeks 24 and 48. Blood and urine sampling to assess the Ca-phosphorous (PO4) axis, parathyroid hormone (PTH)-FGF23-vitamin D signaling, bone turnover, and renal glomerular and tubular function will occur at baseline and study weeks 12, 24, and 48. Blood samples to measure Gluc homeostasis will be drawn at baseline and week 48, and will be run by batch analysis.

Safety, measured by serum calcium (SCa) and serum creatinine (SCr), will be monitored by subject's record review at study sites since these labs will generally be measured as a part of routine clinical care. The Adolescent Medicine Trials Network for HIV/AIDS Interventions 109 (ATN 109) study will use the SCa and SCr values obtained within 10 weeks at the time of the visit beginning at the baseline visit. If these evaluations were not performed within the prior 10 weeks they will be drawn at the time of each visit. Viral load and cluster of differentiation 4 (CD4) cell count results will be recorded for this study, ATN 109, at screening, baseline and study weeks 12, 24, 48, and Post-Week 48 provided the evaluations were done within the protocol specified timeframe. If the evaluations were not performed within the protocol specified timeframes they will be drawn at the time of the visit.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrollment, an individual must meet the criteria listed below at the time of randomization:

NOTE: If the DXA scan is scheduled prior to randomization, all eligibility criteria must be met prior to performing the DXA scan.

* Age 16 years and 0 days to 24 years and 364 days;
* Behaviorally infected with HIV (e.g., sexual contact, injection drug use; not infected by perinatal transmission, blood transfusion, or at age younger than 9 years);
* HIV-1 infection as documented in subject's medical record by at least one of the following criteria:

  * reactive HIV screening test result with an antibody based FDA-licensed assay followed by a positive supplemental assay (e.g., HIV-1 Western Blot, HIV-1 Indirect Immunofluorescence, Antibody Differentiation Assay (Multispot)); or
  * positive HIV-1 DNA polymerase chain reaction (PCR) assay; or
  * plasma HIV-1 quantitative RNA assay >1,000 copies/mL; or
  * positive plasma HIV-1 RNA qualitative assay
* Subjects must have at least one documented HIV viral load that is below 200 copies/mL collected following initiation of TDF containing cART and greater than 90 days prior to randomization; no HIV viral load above 200 copies/mL if measured within the 90 days prior to randomization; and an HIV viral load obtained at screening that is below 200 copies/mL.
* Currently being treated for at least 180 days by the time of randomization with a TDF containing cART with at least 2 other FDA approved ARVs (NOTE: This may include a TDF-containing fixed drug combination medication);
* Negative serum hepatitis B surface antigen (HBsAg) at screening or by history within 4 weeks prior to screening (see section 7.1.3);
* Willingness and ability to remain on the same cART regimen for the duration of study participation;
* Willingness and ability to participate in the study, follow all study procedures for the duration of study participation, and provide written informed consent or assent with parental permission, if applicable; and
* For females of child-bearing potential, agreement to use a minimum of one proven-effective method of birth control and willingness to postpone pregnancy for the duration of study participation (see section 5.3.2 for permitted hormonal contraceptives)

Exclusion Criteria:

To be considered eligible for enrollment, an individual must not meet any of the criteria listed below at the time of randomization:

NOTE: If the DXA scan is scheduled prior to randomization, all eligibility criteria must be met prior to performing the DXA scan.

* Prior hypersensitivity to vitamin D;
* History of sarcoidosis, arteriosclerosis, renal stones, glomerulonephritis, interstitial kidney disease, nephrotic syndrome, hypercalcemia, osteoporosis and/or other bone diseases, clinical diagnosis of hypoparathyroidism or hyperparathyroidism;
* Lactation or pregnancy currently or within the past 24 weeks;
* Chemotherapy or radiation therapy for malignancy within the past 12 months;
* Known presence of GI disease that, in the opinion of the clinician, would interfere with study agent administration or absorption (e.g. Crohn's, Colitis);
* For subjects ≥ 18 years, confirmed creatinine clearance < 70 ml/min (estimated glomerular filtration rate (GFR) from SCr using Cockcroft and Gault (CG) equation) and for subjects <18 years, confirmed creatinine clearance < 70ml/min/1.73m2 (estimated GFR from SCr using Schwartz formula (see section 3.5). (Estimated GFR may be calculated using the formulae programmed on the ATN website);
* SCa > Upper Limit Normal (ULN) for local laboratory values (see section 7.1.3);
* Active Grade 3 or higher clinical or laboratory toxicity except atazanavir (ATV) associated indirect hyperbilirubinemia (see section 9.5.2.2);
* Weight is > 350 pounds (lbs) or 159 kilograms (kgs);
* Positive hepatitis C antibody by history or at screening (see section 7.1.3); and
* Use of any medications as specified in sections 5.3.1, 5.3.3 and 5.4.
* Females Only: Use of certain hormonal contraceptives as specified in the protocol.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Havens, MD, Study Chair — MACC Fund Research Center
Locations (17):
- United States (16):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - University of Southern California - NICHD Westat Site, Los Angeles, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center - NICHD Westat Site, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital and the CORE Center, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Johns Hopkins University - NICHD Westat Site, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Institute, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
- San Juan City Hospital (Puerto Rico) - NICHD Westat Site, San Juan, Puerto Rico

REFERENCES:
- [Result] Havens PL, Stephensen CB, Van Loan MD, Schuster GU, Woodhouse LR, Flynn PM, Gordon CM, Pan CG, Rutledge B, Harris DR, Price G, Baker A, Meyer WA 3rd, Wilson CM, Hazra R, Kapogiannis BG, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 109 Study Team. Vitamin D3 Supplementation Increases Spine Bone Mineral Density in Adolescents and Young Adults With Human Immunodeficiency Virus Infection Being Treated With Tenofovir Disoproxil Fumarate: A Randomized, Placebo-Controlled Trial. Clin Infect Dis. 2018 Jan 6;66(2):220-228. doi: 10.1093/cid/cix753. PMID 29020329
- [Derived] Havens PL, Long D, Schuster GU, Gordon CM, Price G, Wilson CM, Kapogiannis BG, Mulligan K, Stephensen CB; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 117 and 109 study teams. Tenofovir disoproxil fumarate appears to disrupt the relationship of vitamin D and parathyroid hormone. Antivir Ther. 2018;23(7):623-628. doi: 10.3851/IMP3269. Epub 2018 Sep 27. PMID 30260797
- See also: ATN website — http://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This research was conducted at 17 clinical sites, with accrual opening 10/2012. Due to budgetary constraints, accrual to protocol Version 1.0 was placed on hold 9/1/2013; follow-up visits for subjects on study continued while accrual was on hold. Version 2.0 opened to accrual on 2/2/2015. The study was closed to accrual on 6/3/1015.
Period: Overall Study
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Started | 109 | 105
Completed | 98 | 87
Not Completed | 11 | 18
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Starting hormone therapy | 1 | 0
Not completed — Missed 4 or more consecutive DOT visits | 2 | 3
Not completed — Inadvertent enrollment | 1 | 1
Not completed — Moved out of the area | 1 | 5
Not completed — Inability to attend required visits | 0 | 1
Not completed — Off study due to multiple obligations | 0 | 1
Not completed — Fails to comply with study requirements | 0 | 1
Not completed — Childcare issues | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants randomized to Group A or Group B who received the intervention, with the exception of two participants (one in each group) who were later determined to have been inadvertent enrollments who did not meet eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo | Total
Number analyzed (Participants) | 108 | 104 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.84 (1.95) | 21.85 (1.55) | 21.84 (1.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 90 | 89 | 179
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 78 | 79 | 157
  Race: Non-black | 30 | 25 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 21 | 24 | 45
  Ethnicity: Non-Hispanic or Non-Latino | 87 | 79 | 166
  Ethnicity: Unknown/Not reported | 0 | 1 | 1
Season Enrolled [Count of Participants; unit: Participants]
  Winter | 44 | 39 | 83
  Spring | 43 | 42 | 85
  Summer | 15 | 18 | 33
  Fall | 6 | 5 | 11
Lumbar spine bone mineral density (BMD) [Median (Inter-Quartile Range); unit: g/cm^2] | 1.06 [0.99 to 1.19] | 1.08 [0.98 to 1.20] | 1.07 [0.99 to 1.19]
Lumbar spine BMD (L1-L4) (Z-score) [Median (Inter-Quartile Range); unit: z-score] — The Z-score is the standard deviation around mean bone mineral density in the lumbar spine, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected to be seen in healthy populations. A negative Z-score indicates lower than average bone mineral density. Low bone mineral density is a frequent finding in HIV-infected individuals, including adolescents and young adults.
  z-score | -0.65 [-1.40 to 0.00] | -0.70 [-1.60 to 0.20] | -0.70 [-1.50 to 0.10]
Total Hip BMD [Median (Inter-Quartile Range); unit: g/cm^2] — Population: Subjects with valid DXA data for Total Hip
  g/cm^2
    number analyzed (Participants) | 107 | 104 | 211
    (all) | 1.06 [0.95 to 1.16] | 1.05 [0.95 to 1.17] | 1.06 [0.95 to 1.17]
Total hip BMD (Z-score) [Median (Inter-Quartile Range); unit: Z-score] — The Z-score is the standard deviation around mean bone mineral density in the total hip, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected to be seen in healthy populations. A negative Z-score indicates lower than average bone mineral density. Low bone mineral density is a frequent finding in HIV-infected individuals, including adolescents and young adults. Population: Subjects with Total hip BMD z-score data
  Z-score
    number analyzed (Participants) | 105 | 104 | 209
    (all) | -0.40 [-1.10 to 0.10] | -0.65 [-1.35 to 0.00] | -0.50 [-1.20 to 0.00]
Femoral neck BMD [Median (Inter-Quartile Range); unit: g/cm^2] — Population: Subjects with valid DXA data for Femoral Neck
  g/cm^2
    number analyzed (Participants) | 107 | 104 | 211
    (all) | 0.98 [0.88 to 1.12] | 1.00 [0.88 to 1.12] | 0.99 [0.88 to 1.12]
Femoral neck BMD (Z-score) [Median (Inter-Quartile Range); unit: Z-score] — The Z-score is the standard deviation around mean bone mineral density in the femoral neck, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected to be seen in healthy populations. A negative Z-score indicates lower than average bone mineral density. Low bone mineral density is a frequent finding in HIV-infected individuals, including adolescents and young adults. Population: Subjects with available Femoral Neck z-score for baseline
  Z-score
    number analyzed (Participants) | 105 | 104 | 209
    (all) | -0.50 [-1.20 to 0.30] | -0.60 [-1.30 to 0.25] | -0.60 [-1.20 to 0.30]
Whole Body BMD [Median (Inter-Quartile Range); unit: g/cm^2] | 1.18 [1.10 to 1.25] | 1.17 [1.07 to 1.26] | 1.17 [1.09 to 1.25]
Whole body BMD (Z-score) [Median (Inter-Quartile Range); unit: Z-score] — The Z-score is the standard deviation around mean bone mineral density in the whole body, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected to be seen in healthy populations. A negative Z-score indicates lower than average bone mineral density. Low bone mineral density is a frequent finding in HIV-infected individuals, including adolescents and young adults.
  Z-score | -0.60 [-1.35 to 0.10] | -0.80 [-1.65 to 0.10] | -0.70 [-1.60 to 0.10]
Whole Body Bone Mineral Content (BMC) [Median (Inter-Quartile Range); unit: g] | 2636.03 [2368.41 to 2938.59] | 2596.06 [2316.00 to 2936.00] | 2627.16 [2338.39 to 2938.59]
Serum Calcium (SCa) [Median (Inter-Quartile Range); unit: mg/dL] | 9.40 [9.22 to 9.58] | 9.34 [9.14 to 9.58] | 9.39 [9.16 to 9.58]
Urinary Calcium/ Urinary Creatinine ratio (UCa/UCr) [Median (Inter-Quartile Range); unit: ratio] — Population: Subjects with Uca/Ucr lab data available
  ratio
    number analyzed (Participants) | 107 | 103 | 210
    (all) | 0.04 [0.02 to 0.07] | 0.04 [0.02 to 0.07] | 0.04 [0.02 to 0.07]
Serum Phosphate (SPO4) [Median (Inter-Quartile Range); unit: mg/dL] | 3.56 [3.25 to 3.87] | 3.50 [3.19 to 3.86] | 3.52 [3.22 to 3.86]
Tubular reabsorption of phosphate (TRP) % [Median (Inter-Quartile Range); unit: percent] — Population: Subjects with TRP % lab data available
  percent
    number analyzed (Participants) | 107 | 103 | 210
    (all) | 91.72 [89.16 to 93.84] | 91.53 [88.76 to 94.16] | 91.56 [88.91 to 93.94]
Vitamin D serum concentration (25-(OH)D Total) [Median (Inter-Quartile Range); unit: ng/mL] | 15.69 [12.14 to 24.89] | 16.76 [10.18 to 22.68] | 16.37 [11.36 to 23.85]
C-terminal telopeptides (CTX) [Median (Inter-Quartile Range); unit: mcg/L] | 0.76 [0.56 to 1.10] | 0.78 [0.59 to 1.08] | 0.77 [0.58 to 1.09]
Parathyroid hormone (PTH) [Median (Inter-Quartile Range); unit: pg/mL] — Population: Subjects with available data
  pg/mL
    number analyzed (Participants) | 107 | 103 | 210
    (all) | 38.72 [28.81 to 48.52] | 37.04 [28.74 to 46.55] | 37.73 [28.81 to 47.43]
Fibroblast growth factor 23 (FGF23) [Median (Inter-Quartile Range); unit: pg/mL] | 33.23 [26.70 to 42.68] | 34.53 [27.00 to 42.07] | 33.99 [26.72 to 42.57]
Serum 125 dihydroxy vitamin D (125-OHD) [Median (Inter-Quartile Range); unit: pg/mL] — Population: Subjects with available data
  pg/mL
    number analyzed (Participants) | 107 | 104 | 211
    (all) | 72.54 [58.32 to 89.53] | 68.94 [57.13 to 96.09] | 71.08 [57.86 to 93.05]
Actual Free 125(OH)D [Median (Inter-Quartile Range); unit: fmol/L] — Vitamin D serum concentration (1,25 (OH)DTotal) (pmol/L) multiplied by F times 1,000, where F is defined as F = 1/(1 + Kd * [VDBP] + Ka *[albumin]) where the binding constant for vitamin D binding protein (VDBP) = Kd = 4.2 x 107 M-1, and for albumin is Ka = 5.4 x 104 M-1 and the concentrations of VDBP and albumin are in moles/L Population: Subjects with available data
  fmol/L
    number analyzed (Participants) | 107 | 104 | 211
    (all) | 418.48 [315.19 to 638.04] | 445.29 [311.85 to 638.18] | 422.91 [315.19 to 638.04]
Serum Creatinine (SCr) [Median (Inter-Quartile Range); unit: mg/dL] | 0.89 [0.76 to 0.99] | 0.86 [0.76 to 0.96] | 0.86 [0.76 to 0.98]
Estimated glomerular filtration rate (eGFR) [Median (Inter-Quartile Range); unit: ml/min/1.73m^2] — Calculated by the chronic kidney disease (CKD)-Epi equation for subjects > =18 years of age; and by bedside Schwartz formula for subjects <18 years of age
  ml/min/1.73m^2 | 125.02 [114.15 to 140.02] | 125.62 [112.82 to 142.16] | 125.03 [112.82 to 141.01]
Urine Glucose (UGluc) [Median (Inter-Quartile Range); unit: mg/dL] | 7.16 [5.13 to 9.35] | 7.40 [5.46 to 11.26] | 7.27 [5.34 to 10.08]
Urine retinol binding protein (URBP)/ Urine creatinine (UCr) [Median (Inter-Quartile Range); unit: mcg/g] — Population: Subjects with available data
  mcg/g
    number analyzed (Participants) | 107 | 102 | 209
    (all) | 101.21 [70.14 to 142.45] | 104.00 [75.93 to 163.08] | 101.21 [71.63 to 146.62]
Urine beta-2 microglobulin (UB2MG) [Median (Inter-Quartile Range); unit: mcg/L] — Population: Subjects with available data
  mcg/L
    number analyzed (Participants) | 107 | 101 | 208
    (all) | 111.17 [53.28 to 389.38] | 134.08 [51.91 to 305.93] | 127.95 [52.59 to 348.24]
Urine protein (UProt) / Urine creatinine (UCr) [Median (Inter-Quartile Range); unit: ratio] — Population: Subjects with available data
  ratio
    number analyzed (Participants) | 107 | 103 | 210
    (all) | 0.07 [0.05 to 0.08] | 0.07 [0.05 to 0.09] | 0.07 [0.05 to 0.09]
Bone specific alkaline phosphatase (BAP) [Median (Inter-Quartile Range); unit: U/L] | 31.49 [25.28 to 36.74] | 31.76 [25.41 to 37.94] | 31.62 [25.51 to 37.69]
Osteocalcin (OC) [Median (Inter-Quartile Range); unit: mcg/L] | 9.60 [6.47 to 11.63] | 8.94 [5.97 to 11.82] | 9.21 [6.20 to 11.67]
Glucose Homeostasis (Fasting insulin) [Median (Inter-Quartile Range); unit: uIU/mL] — Population: Subjects with available data
  uIU/mL
    number analyzed (Participants) | 108 | 103 | 211
    (all) | 8.87 [5.57 to 12.39] | 8.69 [6.05 to 14.89] | 8.70 [5.59 to 13.82]
Glucose Homeostasis (Fasting glucose) [Median (Inter-Quartile Range); unit: mg/dL] — Population: Subjects with available data
  mg/dL
    number analyzed (Participants) | 107 | 103 | 210
    (all) | 85.55 [81.15 to 91.45] | 86.55 [81.05 to 91.10] | 85.68 [81.05 to 91.25]
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) [Median (Inter-Quartile Range); unit: units on a scale] — Calculated as fasting glucose (mg/dL) X fasting insulin (uIU/mL) /405 Population: Subjects with available data
  units on a scale
    number analyzed (Participants) | 107 | 102 | 209
    (all) | 1.86 [1.07 to 2.65] | 1.78 [1.26 to 3.09] | 1.85 [1.19 to 2.98]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 48 in Dual Energy X-ray Absorptiometry (DXA)-Measured BMD at the Spine for the Randomized Study Groups
Description: Percent change from baseline to week (wk) 48 in DXA-measured BMD at the spine for the randomized study groups.
  Lumbar spine BMD (L1 - L4) (g/cm2) change from Baseline to wk 48 visit.
Time Frame: Baseline and wk 48
Population: Subjects who had baseline and wk 48 data. This includes subjects enrolled in v1.0, who completed wk 48 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be greater than the number completed in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 89
percent change | 0.19 [-1.54 to 1.48] | 0.09 [-1.49 to 2.61]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test type: Other; p = 0.1166, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon rank sum test for change between baseline and Week 48 Vitamin D vs. Placebo

2. Secondary Outcome: Percent Change From Baseline to Week 24 of BMC of Whole Body for the Randomized Study Groups
Time Frame: Baseline and week 24
Population: Subjects who had baseline and wk 24 data. This includes subjects enrolled in v1.0, who completed wk 24 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be greater than the number completed in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
percent change | 0.25 [-1.23 to 1.44] | 0.07 [-0.82 to 1.09]

3. Secondary Outcome: Percent Change From Baseline to Week 48 of BMC of Whole Body for the Randomized Study Groups
Time Frame: Baseline and week 48
Population: Subjects who had baseline and wk 48 data. This includes subjects enrolled in v1.0, who completed wk 48 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the number completed in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 89
percent change | 0.08 [-1.47 to 1.47] | 0.07 [-1.47 to 0.98]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.8383, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percent Change From Baseline to Week 24 of Lumbar Spine (L1-L4) BMD for the Randomized Study Groups
Time Frame: Baseline and week 24
Population: Subjects who had baseline and wk 24 data. This includes subjects enrolled in v1.0, who completed wk 24 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the number completed in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
percent change | 0.94 [-0.72 to 2.16] | 0.42 [-1.02 to 1.91]

5. Secondary Outcome: Change From Baseline to Week 24 of Lumbar Spine (L1-L4) BMD Z-score for the Randomized Study Groups
Description: The Z-score is the standard deviation around mean bone mineral density in the lumbar spine, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected to be seen in healthy populations. A negative Z-score indicates lower than average bone mineral density. Low bone mineral density is a frequent finding in HIV-infected individuals, including adolescents and young adults.
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
z-score | 0.00 [-0.10 to 0.20] | 0.00 [-0.10 to 0.10]

6. Secondary Outcome: Change From Baseline to Week 48 of Lumbar Spine (L1-L4) BMD Z-score for the Randomized Study Groups
Description: as for outcome 5
Time Frame: Baseline and week 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 89
z-score | 0.00 [-0.10 to 0.10] | -0.10 [-0.30 to 0.20]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.1378, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percent Change From Baseline to Week 24 of Femoral Neck BMD for the Randomized Study Groups
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
percent change | -0.10 [-2.49 to 1.65] | -0.04 [-2.16 to 2.13]

8. Secondary Outcome: Percent Change From Baseline to Week 48 of Femoral Neck BMD for the Randomized Study Groups
Time Frame: Baseline and week 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 89
percent change | -0.30 [-2.63 to 1.73] | -0.11 [-2.45 to 1.96]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.4686, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline to Week 24 of Femoral Neck BMD Z-score for the Randomized Study Groups
Description: The Z-score is the standard deviation around mean bone mineral density in the femoral neck, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected to be seen in healthy populations. A negative Z-score indicates lower than average bone mineral density. Low bone mineral density is a frequent finding in HIV-infected individuals, including adolescents and young adults.
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
z-score | 0.00 [-0.20 to 0.10] | 0.00 [-0.10 to 0.20]

10. Secondary Outcome: Change From Baseline to Week 48 of Femoral Neck BMD Z-score for the Randomized Study Groups
Description: as for outcome 9
Time Frame: Baseline and week 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 97 | 89
z-score | 0.00 [-0.20 to 0.10] | 0.00 [-0.20 to 0.10]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.7601, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Percent Change From Baseline to Week 24 of Total Hip BMD for the Randomized Study Groups
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
percent change | -0.27 [-1.08 to 1.53] | 0.00 [-1.14 to 1.46]

12. Secondary Outcome: Percent Change From Baseline to Week 48 of Total Hip BMD for the Randomized Study Groups
Time Frame: Baseline and week 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 89
percent change | -0.17 [-2.12 to 1.73] | -0.42 [-1.66 to 0.71]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.3978, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change From Baseline to Week 24 of Total Hip BMD Z-score for the Randomized Study Groups
Description: The Z-score is the standard deviation around mean bone mineral density in the total hip, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected to be seen in healthy populations. A negative Z-score indicates lower than average bone mineral density. Low bone mineral density is a frequent finding in HIV-infected individuals, including adolescents and young adults.
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 101 | 98
z-score | 0.00 [-0.10 to 0.10] | 0.00 [-0.10 to 0.10]

14. Secondary Outcome: Change From Baseline to Week 48 of Total Hip BMD Z-score for the Randomized Study Groups
Description: as for outcome 13
Time Frame: Baseline and week 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 97 | 89
z-score | 0.00 [-0.10 to 0.10] | 0.00 [-0.10 to 0.10]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.1187, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change in SCr From Baseline to Week 12.
Description: To assess renal glomerular safety by measuring change in SCr from baseline to week 12 by randomized study group;
Time Frame: Baseline and week 12
Population: Subjects who had baseline and wk 12 data. This includes subjects enrolled in v1.0, who completed wk 12 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the numbers in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
mg/dL | 0.03 [-0.03 to 0.08] | 0.02 [-0.03 to 0.07]

16. Secondary Outcome: Change in SCr From Baseline to Week 24.
Description: To assess renal glomerular safety by measuring change in SCr from baseline to week 24 by randomized study group;
Time Frame: Baseline and week 24
Population: Subjects who had baseline and wk 24 data. This includes subjects enrolled in v1.0, who completed wk 24 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the numbers in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
mg/dL | 0.02 [-0.03 to 0.08] | 0.02 [-0.04 to 0.06]

17. Secondary Outcome: Change in SCr From Baseline to Week 48.
Description: To assess renal glomerular safety by measuring change in SCr from baseline to week 48 by randomized study group;
Time Frame: Baseline and week 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
mg/dL | 0.03 [-0.02 to 0.08] | 0.01 [-0.03 to 0.07]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.5098, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Change From Baseline to Week 48 in Glucose Homeostasis (Fasting Insulin)
Time Frame: Baseline and 48 weeks
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: uIU/mL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 89
uIU/mL | 0.45 [-2.21 to 3.48] | -0.83 [-3.02 to 3.43]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.2550, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Change From Baseline to Week 48 in Glucose Homeostasis (Fasting Glucose)
Time Frame: Baseline and week 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 90
mg/dL | 0.05 [-5.05 to 4.20] | -0.20 [-4.85 to 3.85]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.6499, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change From Baseline to Week 48 in Glucose Homeostasis (Homeostasis Model Assessment of Insulin Resistance (HOMA-IR))
Description: HOMA-IR is calculated as fasting glucose (mg/dL) X fasting glucose (uIU/mL) / 405. An increase in HOMA-IR means that an individual has become more resistant (less sensitive) to the effects of insulin and thus would be a negative outcome. A reduction in HOMA-IR means that an individual has become more sensitive to the effects of insulin and would be considered a positive outcome.There are no set minimum or maximum scores for HOMA-IR, since it is based on measurements of insulin and glucose, the assays for which may vary. Several studies suggest a cut-off of >2 for any insulin resistance, but "normal" values appear to vary greatly by population (https://www.mdcalc.com/homa-ir-homeostatic-model-assessment-insulin-resistance).
Time Frame: Baseline and week 48
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 98 | 88
units on a scale | 0.07 [-0.56 to 0.82] | -0.15 [-0.80 to 0.83]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.2348, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Change From Baseline to Week 12 in Serum Calcium (SCa)
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
mg/dL | -0.02 [-0.26 to 0.20] | 0.08 [-0.14 to 0.25]

22. Secondary Outcome: Change From Baseline to Week 24 in Serum Calcium (SCa)
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
mg/dL | -0.04 [-0.26 to 0.16] | 0.08 [-0.16 to 0.30]

23. Secondary Outcome: Change From Baseline to Week 48 in Serum Calcium (SCa)
Time Frame: Baseline and wk 48
Population: Subjects who had baseline and wk 48 data. This includes subjects enrolled in v1.0, who completed wk 48 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the numbers in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
mg/dL | 0.00 [-0.22 to 0.25] | 0.04 [-0.12 to 0.26]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.2648, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Change From Baseline to Week 12 in CTX
Time Frame: Baseline and week 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
mcg/L | -0.03 [-0.21 to 0.13] | -0.02 [-0.19 to 0.15]

25. Secondary Outcome: Change From Baseline to Week 24 in CTX
Time Frame: Baseline and week 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
mcg/L | -0.03 [-0.24 to 0.18] | -0.02 [-0.16 to 0.15]

26. Secondary Outcome: Change From Baseline to Week 48 in CTX
Time Frame: Baseline and week 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 91
mcg/L | -0.08 [-0.25 to 0.10] | -0.09 [-0.27 to 0.02]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.3728, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Change From Baseline to Week 12 in OC
Time Frame: Baseline and week 12
Population: Subjects who had baseline and wk 12 data. This includes subjects enrolled in v1.0, who completed wk 12 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the number completed in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
mcg/L | 0.15 [-0.78 to 1.67] | -0.10 [-1.15 to 1.66]

28. Secondary Outcome: Change From Baseline to Week 24 in OC
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
mcg/L | 0.09 [-1.06 to 1.46] | -0.22 [-1.43 to 1.12]

29. Secondary Outcome: Change From Baseline to Week 48 in OC
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 90
mcg/L | -0.93 [-2.10 to 0.62] | -0.48 [-1.95 to 0.41]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.7825, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Change From Baseline to Week 12 in BAP
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
U/L | -1.05 [-4.33 to 1.85] | -1.74 [-3.82 to 0.88]

31. Secondary Outcome: Change From Baseline to Week 24 in BAP
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
U/L | -2.54 [-5.31 to 0.07] | -2.03 [-4.50 to 0.35]

32. Secondary Outcome: Change From Baseline to Week 48 in BAP
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
U/L | -2.71 [-6.44 to -0.51] | -2.19 [-5.58 to 1.06]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.1950, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: Change From Baseline to Week 12 in FGF23
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
pg/ML | 3.31 [-2.99 to 9.21] | 3.90 [-2.28 to 9.21]

34. Secondary Outcome: Change From Baseline to Week 24 in FGF23
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
pg/ML | 2.93 [-4.07 to 8.35] | 3.65 [-4.45 to 10.53]

35. Secondary Outcome: Change From Baseline to Week 48 in FGF23
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
pg/ML | 4.77 [-2.78 to 10.31] | 3.15 [-3.75 to 10.15]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.7127, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Change From Baseline to Week 12 in PTH
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 105 | 99
pg/ML | -2.17 [-10.26 to 4.00] | -0.82 [-7.79 to 3.95]

37. Secondary Outcome: Change From Baseline to Week 24 in PTH
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 101 | 96
pg/ML | -0.25 [-10.38 to 6.70] | -1.71 [-7.78 to 5.65]

38. Secondary Outcome: Change From Baseline to Week 48 in PTH
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 98 | 89
pg/ML | -2.21 [-10.13 to 4.25] | -0.96 [-9.28 to 4.93]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.4676, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Change From Baseline to Week 12 in Actual Free 1,25-OHD
Description: Vitamin D serum concentration (1,25 (OH)DTotal) (pmol/L) multiplied by F times 1,000, where F is defined as F = 1/(1 + Kd * [VDBP] + Ka *[albumin]) where the binding constant for VDBP = Kd = 4.2 x 107 M-1, and for albumin is Ka = 5.4 x 104 M-1 and the concentrations of VDBP and albumin are in moles/L
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: fmol/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 105 | 99
fmol/L | 106.50 [-12.50 to 222.13] | 53.23 [-28.51 to 148.88]

40. Secondary Outcome: Change From Baseline to Week 24 in Actual Free 1,25-OHD
Description: as for outcome 39
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: fmol/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 101 | 98
fmol/L | 98.61 [-29.77 to 242.62] | 59.36 [-41.94 to 162.45]

41. Secondary Outcome: Change From Baseline to Week 48 in Actual Free 1,25-OHD
Description: as for outcome 39
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: fmol/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 91
fmol/L | 63.73 [-19.39 to 202.54] | 25.66 [-100.82 to 118.45]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.0210, Wilcoxon (Mann-Whitney)

42. Secondary Outcome: Change From Baseline to Week 12 in 1,25-OHD
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 105 | 100
pg/ML | 15.61 [-0.32 to 35.18] | 6.06 [-7.63 to 25.52]

43. Secondary Outcome: Change From Baseline to Week 24 in 1,25-OHD
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 102 | 98
pg/ML | 12.90 [-7.57 to 36.58] | 8.58 [-8.96 to 27.02]

44. Secondary Outcome: Change From Baseline to Week 48 in 1,25-OHD
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: pg/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 99 | 91
pg/ML | 10.52 [-2.05 to 31.47] | 2.74 [-14.73 to 24.48]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.0144, Wilcoxon (Mann-Whitney)

45. Secondary Outcome: Change From Baseline to Week 12 in 25-OHD
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: ng/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
ng/ML | 16.33 [9.33 to 21.19] | 6.91 [2.34 to 11.55]

46. Secondary Outcome: Change From Baseline to Week 24 in 25-OHD
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: ng/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
ng/ML | 18.60 [10.53 to 25.58] | 6.78 [1.35 to 11.24]

47. Secondary Outcome: Change From Baseline to Week 48 in 25-OHD
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: ng/ML
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
ng/ML | 17.80 [11.83 to 24.03] | 2.64 [-1.66 to 7.52]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney)

48. Secondary Outcome: Change From Baseline to Week 12 in TRP %
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 105 | 98
percent | -0.71 [-3.46 to 2.03] | 0.04 [-2.78 to 3.37]

49. Secondary Outcome: Change From Baseline to Week 24 in TRP %
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 101 | 95
percent | -0.59 [-4.43 to 1.79] | -0.88 [-3.001 to 2.32]

50. Secondary Outcome: Change From Baseline to Week 48 in TRP %
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 98 | 87
percent | -1.55 [-4.71 to 1.84] | 0.62 [-2.92 to 3.06]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.0814, Wilcoxon (Mann-Whitney)

51. Secondary Outcome: Change From Baseline to Week 12 in SPO4
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
mg/dL | 0.00 [-0.34 to 0.26] | 0.02 [-0.33 to 0.38]

52. Secondary Outcome: Change From Baseline to Week 24 in SPO4
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
mg/dL | -0.06 [-0.42 to 0.29] | 0.03 [-0.34 to 0.34]

53. Secondary Outcome: Change From Baseline to Week 48 in SPO4
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
mg/dL | -0.03 [-0.33 to 0.36] | -0.12 [-0.47 to 0.31]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.4808, Wilcoxon (Mann-Whitney)

54. Secondary Outcome: Change From Baseline to Week 12 in UCa/Ucr
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 105 | 98
ratio | 0.00 [-0.02 to 0.04] | 0.00 [-0.01 to 0.04]

55. Secondary Outcome: Change From Baseline to Week 24 in UCa/Ucr
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 101 | 95
ratio | 0.01 [-0.01 to 0.05] | 0.01 [-0.01 to 0.02]

56. Secondary Outcome: Change From Baseline to Week 48 in UCa/Ucr
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 98 | 87
ratio | 0.00 [-0.01 to 0.03] | 0.01 [-0.01 to 0.04]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.3870, Wilcoxon (Mann-Whitney)

57. Secondary Outcome: Change in Estimated GFR From Baseline to Week 12.
Description: To assess renal glomerular safety by measuring change in estimated GFR from baseline to week 12 by randomized study group.
  eGFR calculated by the CKD-Epi equation for subjects >=18 years of age, and by bedside Schwartz formula for subjects <18 years of age
Time Frame: Baseline and wk 12
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73m^2
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
ml/min/1.73m^2 | 0.00 [-12.11 to 6.29] | 0.00 [-7.49 to 7.18]

58. Secondary Outcome: Change in Estimated GFR From Baseline to Week 24.
Description: To assess renal glomerular safety by measuring change in estimated GFR from baseline to week 24 by randomized study group;
Time Frame: Baseline and wk 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73m^2
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
ml/min/1.73m^2 | 0.00 [-15.24 to 2.43] | 0.00 [-10.42 to 7.71]

59. Secondary Outcome: Change in Estimated GFR From Baseline to Week 48.
Description: To assess renal glomerular safety by measuring change in estimated GFR from baseline to week 48 by randomized study group;
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73m^2
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
ml/min/1.73m^2 | -1.91 [-15.67 to 3.70] | 0.00 [-10.96 to 5.65]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D) vs. Group B (Placebo); Test type: Other; p = 0.4290, Wilcoxon (Mann-Whitney)

60. Secondary Outcome: Change in UGluc From Baseline to Week 48
Description: To assess renal tubular function by measuring change in urine glucose (UGluc) by randomized study group;
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
mg/dL | -0.42 [-3.27 to 3.23] | -0.43 [-3.17 to 2.62]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.9186, Wilcoxon (Mann-Whitney)

61. Secondary Outcome: Change in URBP/UCr Ratio From Baseline to Week 48
Description: To assess renal tubular function by measuring change in urine retinol binding protein to urine creatinine (URBP/UCr) ratio by randomized study group;
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: mcg/g
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 98 | 88
mcg/g | -1.06 [-37.77 to 32.56] | -4.72 [-33.97 to 18.15]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.4016, Wilcoxon (Mann-Whitney)

62. Secondary Outcome: Change in UB2MG From Baseline to Week 48
Description: To assess renal tubular function by measuring change in urine beta-2 microglobulin (UB2MG) by randomized study group;
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 98 | 89
mcg/L | 5.19 [-95.04 to 111.85] | 10.75 [-90.69 to 157.26]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.5810, Wilcoxon (Mann-Whitney)

63. Secondary Outcome: Change in UProt/ UCr Ratio From Baseline to Week 48
Description: To assess renal tubular function by measuring change in urinary protein to creatinine ratio by randomized study group;
Time Frame: Baseline and wk 48
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 98 | 90
ratio | 0.00 [-0.02 to 0.01] | 0.00 [-0.01 to 0.01]
Statistical Analysis 1: Comparison: Group A: Vitamin D3 50,000 IU vs Group B: Vitamin D3 Placebo; Test for change between baseline and Week 48 Group A (Vitamin D3) vs. Group B (Placebo); Test type: Other; p = 0.1570, Wilcoxon (Mann-Whitney)

64. Secondary Outcome: 25-OHD Serum Concentration by Randomized Study Group at Week 12
Time Frame: Week 12
Population: Subjects who had wk 12 data. This includes subjects enrolled in v1.0, who completed wk 12 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the numbers in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 106 | 100
ng/mL | 35.14 [29.79 to 39.76] | 23.97 [18.35 to 30.19]

65. Secondary Outcome: 25-OHD Serum Concentration by Randomized Study Group at Week 24
Time Frame: Week 24
Population: Subjects who had wk 24 data. This includes subjects enrolled in v1.0, who completed wk 24 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the numbers in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 103 | 98
ng/mL | 37.04 [30.41 to 44.12] | 23.30 [17.92 to 28.49]

66. Secondary Outcome: 25-OHD Serum Concentration by Randomized Study Group at Week 48
Time Frame: Week 48
Population: Subjects who had wk 48 data. This includes subjects enrolled in v1.0, who completed wk 48 evaluations, but were prematurely discontinued before the wk 96 or Post-wk 48 visits and therefore not counted as having completed the study. Thus, the number analyzed may be different from the numbers in the Participant Flow section.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
Number analyzed (Participants) | 100 | 91
ng/mL | 36.89 [30.46 to 42.38] | 20.55 [14.35 to 25.80]

67. Secondary Outcome: Effect of Concurrent Treatment With Efavirenz on 25-OHD Serum Concentration: Concentration at Baseline by Efavirenz Use
Description: Mean Vitamin D serum concentration (25-(OH)D) Total) in those with efavirenz use vs. those without efavirenz use
Time Frame: Baseline
Population: Authors were interested in comparing mean 25-OHD at baseline by those who used efavirenz vs those who did not use efavirenz; a separate analysis by treatment arm was not done. Due to different comparison groups, the number of subjects analyzed differ from the numbers in the Participant Flow section.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Efavirenz Use: Ever used efavirenz
- No Efavirenz Use: Never used efavirenz
Arm/Group | Efavirenz Use | No Efavirenz Use
Number analyzed (Participants) | 78 | 134
ng/mL | 17.02 (8.69) | 19.61 (9.96)

68. Secondary Outcome: Effect of Concurrent Treatment With Efavirenz on 25-OHD Serum Concentration: Concentration at Week 48 by Efavirenz Use
Description: Mean Vitamin D serum concentration (25-(OH)D) Total) in those with efavirenz use vs. those without efavirenz use
Time Frame: Week 48
Population: Authors were interested in comparing mean 25-OHD at wk 48 by those who used efavirenz vs those who did not use efavirenz; a separate analysis by treatment arm was not done. Due to different comparison groups, the number of subjects analyzed differ from the numbers in the Participant Flow section.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Efavirenz Use | No Efavirenz Use
Number analyzed (Participants) | 72 | 119
ng/mL | 28.24 (11.22) | 29.68 (11.52)

69. Secondary Outcome: Effect of Concurrent Treatment With Efavirenz on 25-OHD Serum Concentration: Change in Concentration From Baseline to Week 48 by Efavirenz Use
Description: Mean Vitamin D serum concentration (25-(OH)D) Total) in those with efavirenz use vs. those without efavirenz use
Time Frame: Baseline and wk 48
Population: Authors were interested in comparing the change in mean 25-OHD from baseline to wk 48 by those who used efavirenz vs those who did not use efavirenz; a separate analysis by treatment arm was not done. Due to different comparison groups, the number of subjects analyzed differ from the numbers in the Participant Flow section.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Efavirenz Use | No Efavirenz Use
Number analyzed (Participants) | 72 | 119
ng/mL | 10.97 (12.00) | 9.79 (11.68)
Statistical Analysis 1: Comparison: Efavirenz Use; Test of change from baseline to week 48; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: No Efavirenz Use; Test of change from baseline to Week 48; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test

70. Secondary Outcome: Effect of Concurrent Treatment With Ritonavir on 25-OHD Serum Concentration: Concentration at Baseline by Ritonavir Use
Description: Mean Vitamin D serum concentration (25-(OH)D) Total) in those with ritonavir use vs. those without ritonavir use
Time Frame: Baseline
Population: Authors were interested in comparing mean 25-OHD at baseline by those who used ritonavir vs those who did not use ritonavir; a separate analysis by treatment arm was not done. Due to different comparison groups, the number of subjects analyzed differ from the numbers in the Participant Flow section.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ritonavir Use: Ever used ritonavir
- No Ritonavir Use: Never used ritonavir
Arm/Group | Ritonavir Use | No Ritonavir Use
Number analyzed (Participants) | 88 | 124
ng/mL | 18.62 (8.79) | 18.69 (10.13)

71. Secondary Outcome: Effect of Concurrent Treatment With Ritonavir on 25-OHD Serum Concentration: Concentration at Week 48 by Ritonavir Use
Description: Mean Vitamin D serum concentration (25-(OH)D) Total) in those with ritonavir use vs. those without ritonavir use
Time Frame: Week 48
Population: Authors were interested in comparing mean 25-OHD at wk 48 by those who used ritonavir vs those who did not use ritonavir; a separate analysis by treatment arm was not done. Due to different comparison groups, the number of subjects analyzed differ from the numbers in the Participant Flow section.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ritonavir Use | No Ritonavir Use
Number analyzed (Participants) | 77 | 114
ng/mL | 29.46 (10.70) | 28.92 (11.89)

72. Secondary Outcome: Effect of Concurrent Treatment With Ritonavir on 25-OHD Serum Concentration: Change in Concentration From Baseline to Week 48 by Ritonavir Use
Description: Mean Vitamin D serum concentration (25-(OH)D) Total) in those with ritonavir use vs. those without ritonavir use
Time Frame: Baseline and wk 48
Population: Authors were interested in comparing the change in mean 25-OHD from baseline to wk 48 by those who used ritonavir vs those who did not use ritonavir; a separate analysis by treatment arm was not done. Due to different comparison groups, the number of subjects analyzed differ from the numbers in the Participant Flow section.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ritonavir Use | No Ritonavir Use
Number analyzed (Participants) | 77 | 114
ng/mL | 10.55 (11.07) | 10.02 (12.28)
Statistical Analysis 1: Comparison: Ritonavir Use; Test of Week 48 difference from baseline; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: No Ritonavir Use; Test of Week 48 difference from baseline; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test

ADVERSE EVENTS:
Time Frame: Adverse events were collected between Baseline through Week 48 or premature discontinuation from study.
Arm/Group | Group A: Vitamin D3 50,000 IU | Group B: Vitamin D3 Placebo
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/105
Serious Adverse Events (participants affected / at risk) | 5/109 | 6/105
Other Adverse Events (participants affected / at risk) | 6/109 | 8/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Vitamin D3 50,000 IU (N=109) | Group B: Vitamin D3 Placebo (N=105)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Vitamin D3 50,000 IU (N=109) | Group B: Vitamin D3 Placebo (N=105)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1)
Streptococcus Test (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The analysis by efavirenz use and ritonavir use after baseline do not adjust for treatment group (secondary outcome measures 68, 69, 71, and 72). Results post-baseline may differ based on treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications, and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by the protocol team and AMLG.